CLINICAL TRIAL: NCT03193996
Title: 4DCT Imaging for Improved Diagnosis and Treatment of Wrist Ligament Injuries
Acronym: 4DCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristin Zhao, PhD (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Kristin Zhao, PhD, Assistant Professor of Biomedical Engineering, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-001279; 1R01AR071338-01 (NIH)
Record Dates: First submitted 2017-06-15; First posted 2017-06-21 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Scapholunate Interosseous Ligament Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SLIL Injury (Other): Surgical interventions for all subjects will be determined based on combined findings of both 4DCT and standard arthroscopy.
  Interventions: Device: 4DCT

INTERVENTIONS:
Device: 4DCT — 4DCT will be used to assess the location of the torn scapholunate interosseus ligament.

SUMMARY:
The study seeks to determine whether the 4DCT imaging technique can be used to replace current invasive diagnostic tests for ligament injuries of the wrist.

DETAILED DESCRIPTION:
Aim 1:

40 cadaveric forearm/hand specimens will be obtained from the Mayo Clinic Anatomical Bequest program. 10 will be used to refine the ligament injury model and 30 will be used as follows. The specimens will undergo radiographic screening and will be excluded from the study if they have evidence of fracture, bony trauma, significant arthritic changes, or previous surgeries. The tendons will be loaded. The remaining soft tissues will be dissected from the proximal ulna and radius. Polymethylmethacrylate (PMMA) resin will be used to affix the proximal radius and ulna in a circular acrylic fixture. The custom wrist motion simulator was designed to generate muscle-assisted flexion-extension and radial-ulnar deviation movements and is CT-compatible. Each tendon will be dynamically loaded with a constant 10 N, maintained throughout the movement in the following conditions: wrist flexion-extension and radial-ulnar deviation. The hand will be fixed in a grip that is connected to a programmable linear actuator. The linear actuator drives the grip back-and-forth along the x-axis with free-motion along the z-axis. The linear actuator will be programmed to allow the wrist to perform a full radial-ulnar or flexion-extension motion at 30 deg/sec which simulates in vivo wrist motion speeds. A motion cycle is approximately 2 seconds. The wrist will be cycled 100 times in flexion-extension prior to each testing condition. A static CT image will be acquired in the neutral posture. Then, each wrist will be imaged using 4DCT during flexion-extension and radial-ulnar deviation, in the following conditions: intact (control), volar SLIL cut, membranous SLIL cut, dorsal SLIL cut, radioscaphocapitate ligament cut, and long radiolunate ligament cut.

Aim 2:

4DCT scanning will be performed bilaterally on 60 patients (30 males, 30 females) with unilateral SLIL injury who are scheduled to undergo a surgical intervention. In addition, patients will have pre-surgical volar and dorsal arthroscopic confirmation of ligament injury, categorized by Geissler and European Wrist Arthroscopy Society (EWAS) classifications; video recording of the arthroscopy will be obtained for later analysis. PRWE and VAS questionnaires will be completed at the 4DCT visit for the injured wrist and the Total Patient Rated Wrist Evaluation (PRWE) score (sum of pain and function subscales) and composite change in Visual Analog Pain Scale (VAS) score used in the analysis. 4DCT wrist data will be obtained while the subjects perform flexion-extension and radial-ulnar deviation. The dynamic image sequence will be processed with existing software tools to obtain metrics describing the interosseous distances between the articular surfaces of the scaphoid, lunate, and radius, during the movement cycles. Given the difficulty of diagnosing SLIL injury, the uninjured contralateral wrist is often used as a "control" for comparison by physicians; therefore, the difference in right/left metrics will be used in the study.

Aim 3:

The same 60 patients ( see Aim 2) will be evaluated. Surgeons will assess pre-surgical scapholunate interosseus distances (quantified using 4DCT in Aim 2) and document a treatment plan to address the particular injury. Subsequently, 4DCT-based treatment plans will be compared with arthroscopic evaluation (obtained in Aim 2); any existing wrist x-rays (e.g. AP, lateral, stress views) and MRIs may be used in this comparison as well. The surgeon will then select and perform the targeted surgical intervention based on both 4DCT and arthroscopic findings. 4DCT will be performed, and the PRWE and VAS completed by patients at 1 year postoperatively; quantification of radioscaphoid contact patterns will be assessed during bilateral wrist flexion-extension and radial-ulnar deviation to determine if normal patterns of motion are restored.

ELIGIBILITY:
Inclusion Criteria:

1. unilateral scapholunate instability
2. point tenderness over the dorsal aspect of the scapholunate joint
3. positive Watson shift sign (Watson et al., J Hand Surg Am, 1988; 13:657-60);
4. suspected pathology on previous fluoroscopy or MRI;

Exclusion Criteria:

1. previously-diagnosed rheumatological conditions or connective tissue diseases
2. inability to be appropriately positioned in the scanner for the imaging
3. congenital malformations of the wrist or forearm
4. diagnosed wrist osteoarthritis
5. age under 18 or over 60

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin D. Zhao, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SLIL Injury
Started | 29
Completed | 16
Not Completed | 13
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 2
Not completed — Pregnancy | 1
Not completed — Subject did not proceed to reconstructive surgery. | 1
Not completed — Complicating disease | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | SLIL Injury
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Equivalency of 4DCT-based Treatment Plan to Arthroscopic-based Treatment Plan.
Description: Baseline, Post-4DCT Viewing, Post-Arthroscopy estimates or observations were made by the attending surgeon of Geissler grading, an arthroscopic classification of carpal instability and suggested management of acute injuries to the SLIL. Lower Geissler grading indicates milder damage and suggests more conservative injury management, and higher Geissler grading indicates more severe damage and suggests more aggressive injury management.
Time Frame: Baseline, Post-4DCT Viewing, Post-Arthroscopy
Population: All participants who underwent 4DCT scanning were analyzed for suspected change in Geissler grade. A subset of participants who proceeded to arthroscopy were analyzed for grading agreement between arthroscopy and 4DCT scan, and between arthroscopy and clinical suspicion prior to the 4DCT scan occurring.
Measure: Count of Participants; unit: Participants
Arm/Group | SLIL Injury
Number analyzed (Participants) | 22
Participants
  4DCT changed suspected Geissler stage | 5
  Agreement in Geissler stage between arthroscopy and 4DCT.: number analyzed (Participants) | 19
  Agreement in Geissler stage between arthroscopy and 4DCT. | 14
  Agreement in Geissler stage between arthroscopy and clinical suspicion pre-4DCT: number analyzed (Participants) | 19
  Agreement in Geissler stage between arthroscopy and clinical suspicion pre-4DCT | 11

2. Secondary Outcome: Subject Perception of Surgical Outcome
Description: Baseline and one year post-surgery Patient-Rated Wrist Evaluation (PRWE) Score will measure patient perception of change. The PRWE allows patients to rate their levels of wrist pain and disability from 0 to 10, with higher numbers representing more pain and disability, and consists of 2 subscales as well as a total score:
  Pain subscale: contains 5 items each of which is further rated from 0-10. The maximum score in this section is 50 and minimum 0, with a higher score suggesting more severe and frequent pain.
  Function subscale: contains total 10 items. The maximum score in this section is 50 and minimum 0, with a higher score suggesting greater difficulty performing activities of daily living.
  Total score: all subscales together. The maximum score in this section is 100 and minimum 0, with a higher score suggesting more pain and disability overall.
Time Frame: Baseline and 1 Year Post-Surgery
Population: All subjects who completed 1-year follow-up evaluation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SLIL Injury
Number analyzed (Participants) | 16
score on a scale
  Pain domain change between baseline and 1-year post surgery | -12.5 [-18 to -6]
  Functional impairment change between baseline and 1-year post surgery | -4.5 [-7.5 to -2]
  Total PRWE score change between baseline and 1-year post surgery | -20 [-24.3 to -8.5]

ADVERSE EVENTS:
Time Frame: At baseline and 1-year post surgery
Description: Subject participation was limited to two single scanning visits separated by approximately one year; as such, temporal association was limited to during and directly after scanning visits.
Arm/Group | SLIL Injury
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT03193996/Prot_SAP_002.pdf
  • Informed Consent Form (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT03193996/ICF_001.pdf